CLINICAL TRIAL: NCT06222151
Title: Recovering From Bariatric Surgery: the Effects of Early Initiated and Supervised Mobilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/44737
Record Dates: First submitted 2023-12-13; First posted 2024-01-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain, Acute; Postoperative Pain, Chronic; Bariatric Surgery; Mobilization; Physical Activity
Keywords: Pain Coping; Bariatric Surgery; Postoperative Pain; Physical Activity; Mobilization
MeSH Terms: conditions — Pain, Postoperative; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into the intervention or control group. To assess the effect of the two interventions separately and independent of each other and to avoid inequality at the starting point of intervention 1 and 2, the patients will at the starting point be randomized into four different groups: A) Intervention 1/Intervention 2, B) Intervention 1/Control 2, C) Control 1/ Intervention 2 D) Control 1/Control 2 (Figure 1). This procedure will enable evaluation of one intervention group versus one control group who are different at each time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): Participates in intervention 1 and 2
  Interventions: Other: Intervention 1: Mobilization during hospitalization; Other: Intervention 2: Mobilization the first 4 postoperative weeks
- B (Other): Participates in intervention 1, control in intervention 2
  Interventions: Other: Intervention 1: Mobilization during hospitalization; Other: Intervention 2: Mobilization the first 4 postoperative weeks; Other: Control group
- C (Other): Participates in intervention 2, control in intervention 1
  Interventions: Other: Intervention 1: Mobilization during hospitalization; Other: Intervention 2: Mobilization the first 4 postoperative weeks; Other: Control group
- D (Active Comparator): Control in both intervention 1 and 2
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention 1: Mobilization during hospitalization — Surgical ICU Optimal Mobilization Score (SOMS) will be used to initiate early mobilization. SOMS consists of five levels of mobilization reaching from no activity to ambulation. Thirty minutes after PACU-arrival, the patient will be asked to do lower leg exercises. If this is possible, the patient will advance to the next level of mobilization. If not possible, level zero is recorded and the patient rests for another 30 minutes before attempting level one again. This continues until the patient succeeds with level four. Safety criteria for advancing to the next level of mobilization are based on criteria for mobilizing patients in the ICU. The intervention group will receive standard care with additional supervised mobilization while hospitalized. This mobilization consist of walking 1000 steps on postoperative day (POD) 0 and 500 steps on POD1 before discharge. Step counts are measured using pedometers.
  Arms: A; B; C
Other: Intervention 2: Mobilization the first 4 postoperative weeks — Intervention 2 will start the first weekday after discharge and continue for 4 weeks. Four supervised physical activity sessions and 8 sessions using telerehabilitation. The activities are low-intensity exercises (walking and lightly strength training using resistance bands) with progressed intensity throughout the weeks. The exercises will be individually progressed to meet the participant's level of activity, as it is important the participants benefit as much as possible from the intervention. The participants will receive information about different possibilities for leisure activities, for motivation to continue physical activity after the first 4 weeks.
  Arms: A; B; C
Other: Control group — The control group receives standard care.
  Patients are mobilized to sit at the bedside before being transferred to the surgical ward. However, it is not used as prophylactic pain management nor is there a structured evidence based protocol with regard to mobilization. The control group will also be equipped with pedometers. They are encouraged to mobilize, and they receive a form in which they can write down mobilization for each hour. There is no planned supervised mobilization. As patients in the control group are assigned to standard care, they will not receive any supervised physical activity after discharge.
  Arms: B; C; D

SUMMARY:
The aim is to investigate the effect of early initiated and supervised mobilization continued after discharge as management of postoperative pain and recovery following obesity surgery, including patient experiences, pain coping, physical functionality and quality of life.

DETAILED DESCRIPTION:
Study aims;

1. To investigate the effect of mobilization as pain management following obesity surgery.
2. To investigate patient experiences with mobilization and postoperative pain, including the influence of mobilization on patients' ability to cope with pain and an identification of facilitating factors and barriers towards early mobilization.
3. To assess the effect of mobilization on postoperative recovery, including the general physical activity level, physical function, and quality of life among patients discharged after obesity surgery.

The PhD study consists of two sub-studies. Study 1: Effect of early mobilization as pain management in patients recovering from obesity surgery. The study is a single center randomized controlled trial (RCT). Participants will be randomized with an allocation ratio of 1:1.

Study 2: Patient experiences with early mobilization and postoperative pain after surgery - An interview study Patients participating in both interventions (group A), will be invited to participate in two individual semi structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* The ability to read and understand the Danish language

Exclusion Criteria:

* Preoperative dependence of walking aids
* Vision impairment
* Previous syncopes or epilepsy
* Admission to the intensive care unit after surgery
* Acute complications during hospital admission
* Patients are excluded at baseline if they have an oxygen saturation below 90% or a systolic blood pressure above 180 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain | 24 hours post surgery
  Abdominal pain measured using a visual analog scale (VAS) of 0-10. A higher score indicates a worse pain.
Physical function | Baseline, 1 month postoperative and 6 months postoperative
  A 6 minute walk test measured in metres

SECONDARY OUTCOMES:
Abdominal pain | At baseline, during intervention 1, 1 month postoperative and 6 months postoperative
  Abdominal pain measured using a visual analog scale (VAS) of 0-10. A higher score indicates a worse pain.
Morphine equivalent consumption | At baseline, during intervention 1, at discharge (at the end of intervention 1), 1 month postoperative and 6 months postoperative
  Measured in milligram intravenous
Patient reported pain experiences | At baseline, during intervention 1, 1 month postoperative and 6 months postoperative
  APS-POQ-R-D questionnaire.
Pain self-efficacy | At baseline, during intervention 1, 1 month postoperative and 6 months postoperative
  PSEQ-DK questionnaire. Pain self-efficacy is measured on a score of 0-60. A higher score indicates a greater pain self-efficacy.
Pain catastrophizing | At baseline, during intervention 1, 1 month postoperative and 6 months postoperative
  Pain Catastrophizing Scale questionnaire. Pain Catastrophizing is measured on a score of 0-52. A higher score indicates a higher pain catastrophizing.
Postoperative nausea and vomiting | During intervention 1, at discharge (at the end of intervention 1), 1 month postoperative and 6 months postoperative
  On a visual analog scale (VAS) of 0-10. A higher score indicates worse nausea.
Health related quality of life (SF-36) | At baseline, during intervention 1, 1 month postoperative and 6 months postoperative
  Questionnaire SF-36. Health related quality of life is measured at a scale of 0-100. A higher score indicates a greater quality of life.
Physical activity | At baseline, 1 month postoperative and 6 months postoperative
  Measured using accelerometers - minutes low/medium/high activity performed per hour. Measured for 7 days at baseline, 7 days 1 month postoperative and 7 days 7 months postoperative
Readmission | 1 month postoperative and 6 months postoperative
  Readmissions during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Esbjerg Hospital, University Hospital of Southern Denmark, Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen NMN, Oxlund J, Dreyer P, Gram B. Recovery After Bariatric Surgery: The effects of Mobilization-A Study Protocol. Pain Manag Nurs. 2025 Dec 19:S1524-9042(25)00332-7. doi: 10.1016/j.pmn.2025.11.017. Online ahead of print. PMID 41421861